CLINICAL TRIAL: NCT05560243
Title: Development, Implementation, and Evaluation of a Tobacco Cessation Intervention Tailored to Patients Living With HIV (PLWH) in Brazil: A Feasibility Study
Brief Title: Tobacco Cessation Tailored to Patients Living With HIV (PLWH) in Brazil
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: Universidade Estadual de Londrina (Other)
Responsible Party: Principal Investigator, Isabel Scarinci, Professor, University of Alabama at Birmingham
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: R21DA049557 (NIH)
Record Dates: First submitted 2022-09-26; First posted 2022-09-29 (Actual); Results first posted 2024-12-11 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-12

CONDITIONS: HIV Infections; Tobacco Use Cessation
Keywords: HIV, tobacco cessation
MeSH Terms: conditions — HIV Infections; Tobacco Use Cessation | interventions — Tobacco Use Cessation Devices

STUDY DESIGN:
Intervention Model Description: Feasibility of a tobacco cessation program tailored to patients living with HIV
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): Patients will receive a tobacco cessation intervention
  Interventions: Behavioral: Tobacco cessation

INTERVENTIONS:
Behavioral: Tobacco cessation — Tobacco cessation program consisting of cognitive-therapy sessions and pharmacological management

SUMMARY:
The overall goal of this feasibility study is to make adaptations to these evidence-based approaches in collaboration with PLWH and health care providers working with this population, and develop, implement, and evaluate the feasibility and scalability of a theory-based, culturally relevant tobacco cessation intervention for PLWH receiving care through the public health system in a southern town in Brazil (Londrina). This proposal will focus on the intervention development, pretesting, and feasibility testing. The primary outcome will be a 7-day point prevalence abstinence (defined as no tobacco use in the past 7 days and verified through measurement of salivary cotinine and exhaled carbon monoxide levels) at 6-month follow-up. We will also conduct detailed treatment fidelity and scalability assessments (acceptability, feasibility, potential reach and adoption, alignment with the strategic context) to inform a full-scale efficacy trial.

DETAILED DESCRIPTION:
This study aims at developing and examining feasibility and scalability of a theory-based, culturally relevant tobacco cessation intervention for PLWH receiving care through the public health system in a southern town in Brazil. It consists of three phases: formative assessments with patients and health care providers to inform relevant components of the intervention, pretesting of the intervention components, and pilot testing of the intervention (feasibility).

ELIGIBILITY:
Inclusion Criteria:

* PLWH (that is, patients with a confirmed HIV diagnosis) receiving care at the reference center in Londrina
* 18 years of age and older; (c) smoke at least 5 cigarettes (industrialized or hand-rolled) per day Smoked within the past seven days.
* No intent to move from the area served by reference center in Londrina within the next 12 months.

Exclusion Criteria:

* History of hypertension
* History of angina
* History of asthma
* On medication for depression.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2023-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Isabel C Scarinci, PhD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- Universidade Estadual de Londrina, Londrina, Paraná, Brazil

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Intervention
Started | 56 (Although 56 participants consented, only 45 started the intervention.)
Completed | 31
Not Completed | 25
Not completed — 11 did not start the intervention, and 14 were lost to follow-up | 25

BASELINE CHARACTERISTICS:
Arm/Group | Intervention
Number analyzed (Participants) | 45
Age, Continuous [Mean (Standard Deviation); unit: years] | 46 (11.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 28
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Brazil | 45
Educational attainment - completed at least high school [Number; unit: participants] | 25
Number of cigarettes/day [Mean (Standard Deviation); unit: cigarettes/day] | 18.4 (11.4)
Fagerstrom Score - moderate to very high [Number; unit: participants] — Fagerstrom Test for Nicotine Dependence assesses the intensity of physical addiction to nicotine. It contains six items and final score ranges from 0 to 10. Scores between 5 and 10 are considered moderate to very high physical addiction and if of clinical significance.
  participants | 28
Depressive symptomatology (CES-D) [Mean (Standard Deviation); unit: units on a scale] — The Center for Epidemiological Studies Depression Scale (CES-D) assesses self-report depressive symptomatology in the general population. It is a screening test for depressive symptomatology and not a diagnostic test. Scores range from 0 to 60. Scores of 16 and higher are indicative of depressive symptomatology and it requires further assessments. This questionnaire does not have sub-scales.
  units on a scale | 25.8 (15.8)
Social Support [Mean (Standard Deviation); unit: units on a scale] — The Multidimensional Scale of Perceived Social Support assesses the adequacy of social support participants receive. Final scores between 1 and 2.9 indicate low social support, 3-5 moderate social support, and 5-7 high social support.
  units on a scale | 4.5 (1.6)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With a 7-day Prevalence Abstinence of Tobacco Use
Description: 7-day point prevalence abstinence (defined as no tobacco use in the past 7 days and verified through measurement of salivary cotinine and exhaled carbon monoxide (CO) levels) at 6-month follow-up.
Time Frame: 6-month follow-up
Measure: Number; unit: participants
Groups:
- Intervention: Tobacco cessation intervention - pharmacological management and cognitive behavioral therapy
Arm/Group | Intervention
Number analyzed (Participants) | 45
participants | 27

2. Secondary Outcome: Participants With Tobacco Use Abstinence Based on Salivary Cotinine at 7-month Follow-up.
Description: Tobacco use abstinence based on salivary cotinine was assessed at 7-month follow-up
Time Frame: 7 months
Measure: Number; unit: participants
Arm/Group | Intervention
Number analyzed (Participants) | 45
participants | 18

ADVERSE EVENTS:
Time Frame: 12 months
Description: Adverse events were monitored but none reported
Arm/Group | Intervention
All-Cause Mortality (participants affected / at risk) | 0/45
Serious Adverse Events (participants affected / at risk) | 0/45
Other Adverse Events (participants affected / at risk) | 0/45

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-11-20): https://cdn.clinicaltrials.gov/large-docs/43/NCT05560243/Prot_SAP_000.pdf